



## PROCOG TRIAL CONSENT FORM

**Research Study Title: Pro**biotic impact on **Cog**nitive performance, and metabolic outcomes in overweight young adults with impaired glucose regulation (**Pro-Cog**)

## Instructions:

Please read each statement below and tick Yes or No to indicate your agreement. Items 1–15 relate to essential aspects of the study. Items 16–20 are optional; you can still take part in the main study if you choose not to agree to any of the optional items.

| No. | Item | Please tick | |
|---|---|---|---|
| | | Yes | No |
| 1. | I have read and understood the Participant Information Sheet (Version 1.1, Date: 28/08/25). I have had the chance to ask questions, and these have been answered to my satisfaction. | | |
| 2. | I understand that taking part is voluntary and that I can withdraw at any time without giving a reason. | | |
| 3. | I understand that if I withdraw, no further data will be collected. I may ask for my identifiable data to be removed, but anonymised data already collected may still be used. | | |
| 4. | I confirm that I meet the study eligibility criteria as explained to me by the research team. | | |
| 5. | To the best of my knowledge, I am in good health and it is safe for me to take part in this study. I have told the research team about any relevant health conditions or medications. | | |
| 6. | I understand the potential risks of taking part in this study, and these have been explained to me clearly. | | |
| 7. | I understand the potential benefits of taking part in this study, and these have been explained to me clearly. | | |
| 8. | I understand that if a serious health issue is identified during screening, the research team will inform me. In a medical emergency, they may contact emergency services and share only relevant health information as necessary. For non-urgent issues, I am responsible for seeking care from my GP or another provider. | | |
| 9. | I understand that the research team may ask me to stop participating if continuing is no longer in my best interest or if I no longer meet the eligibility criteria. | | |
| 10. | I understand that my personal and research data will be stored securely on Leeds Beckett University systems and handled in line with GDPR and the Data Protection Act 2018. | | |
| 11, | I understand my data will be processed in line with GDPR and UK data protection law. | | |
| 12. | I understand that study findings may be published in scientific journals, shared at conferences, or appear in press releases or on websites, but I will not be personally identifiable. | | |





| 13. | I understand that anonymised data madatabase and shared with other resear students, for secondary analysis, in line ethical standards. | chers, including university | | |
|---|---|---|---|---|
| 14. | I agree to provide blood samples for the analysed for health markers and may be related to this study. | be securely stored for future testing | | |
| 15. | I confirm that the information I have pro<br>and accurate to the best of my knowled | | | |
| | Optional items (you can still take part in the study if you do not agree to these) | | | |
| 16. | I agree to provide stool samples for thi store these samples until my final visit analysed for gut bacteria and may be srelated to this study. | at week 12, and they will be | | |
| 17. | I agree that my anonymised blood and<br>used in future ethically approved resea<br>the microbiome. This may involve univ<br>commercial organisations, in the UK or | arch related to health, probiotics, or ersities, hospitals, non-profits, or | | |
| 18. | I agree to receive reminder messages via text during the study. I understand used for study-related communication Mobile number: | that my phone number will only be | | |
| 19. | I would like to receive the following via email (please tick all that apply): ☐ A summary of overall study findings ☐ My individual results (cognitive performance, body composition, cardiovascular health, | | | |
| Bv siar | ning this consent form, I agree to take p | art in the research study named at th | e top of | f this |
| page. | | | | |
| Name of person giving consent (Please print your name here): Date: Signature: | | Researcher: Lewis Hepburn Date: Signature: | | |